CLINICAL TRIAL: NCT00100412
Title: Cardiovascular Hyporeactivity and Fatiguing Illness in Gulf War Veterans
Brief Title: Hyporeactivity and Gulf War Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Purpose: Diagnostic
Other Study IDs: MHBS-001-99S1
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Gulf War Syndrome; Chronic Fatigue Syndrome; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Persian Gulf Syndrome; Fatigue Syndrome, Chronic; Stress Disorders, Post-Traumatic

INTERVENTIONS:
Drug: Graded dobutamine infusions
Drug: Graded phenylephrine injections
Behavioral: Psychosocial challenge involving socioevaluative public speaking

SUMMARY:
This research project is a follow-up to the prior VA-funded study that found that chronic fatigue reported by many Gulf War veterans may be a symptom of dysfunctional cardiovascular stress response regulation. Specifically, ill veterans had diminished autonomic responses during demanding psychosocial tasks involving high level cognitive processing and emotional stress. There was a close relationship between clinical status of ill veterans and their inability to mount an appropriate physiological response under stress. The main objective of the present investigation is to determine the specific mechanism through which this abnormality may contribute to Gulf War-related chronic fatigue. We also observed that Gulf veterans with posttraumatic stress disorder (PTSD) had the most dampened autonomic activation to stressors involving higher brain activities. The second major focus of this study is to explore the role of a psychiatric disorder, specifically PTSD, as a factor in abnormalities in stress response regulation. This aspect of the study may also provide pertinent information as to the role of stress of military deployment as a contributing factor in post-Gulf War illnesses.

DETAILED DESCRIPTION:
Objective: Our previous VA-funded study found that chronic fatigue reported by some Gulf War veterans may be a symptom of dysfunctional cardiovascular stress response regulation. Specifically, ill veterans had diminished autonomic responses during tasks involving higher brain activities, including cognitive processing and psychosocial stress. Gulf veterans with posttraumatic stress disorder (PTSD) had the most dampened autonomic activation to stressors involving higher brain activities. There was a close relationship between the clinical status of ill veterans and their inability to mount an appropriate physiological response under stress. The main objective of the present investigation is to determine the specific mechanism through which this abnormality may contribute to Gulf War-related chronic fatigue. The second major focus of this study is to explore the role of stress of military deployment as a contributing factor in post-Gulf War illnesses.

Research Plan: The research plan is to establish the mechanisms of blood pressure hyporeactivity in Gulf War veterans with chronic fatigue and PTSD. Two possibilities are being examined: one, that abnormal cardiovascular responses to stressors involve reduced responsiveness of the major cardiovascular effector systems, the peripheral arterial vasculature and the heart, to sympathetic stimulation; and two, that the locus of abnormality is in the brain, resulting in inadequate activation of the sympathetic nervous system during stressful behavioral activities. The role of wartime stress will be examined by specifically focusing on abnormalities in stress response regulation associated with Gulf War-related PTSD.

Methods: This study is being performed on four groups of Gulf War veterans, including those with symptoms that fulfill the 1994 CDC case definition for chronic fatigue syndrome (CFS), those with PTSD, those who have both CFS and PTSD, and healthy control veterans. A total of 90 veterans will be studied. The study protocol uses standard laboratory procedures to characterize abnormalities in regulation of cardiovascular function using selective pharmacological and behavioral challenges. Performance of central mechanisms of sympathetic activation during mental challenge is evaluated by measuring increases in plasma catecholamines, epinephrine and norepinephrine, during social-evaluative speech stressor. Collected plasma samples are analyzed using high performance liquid chromatography assays. The hypotheses of target organ dysfunction are evaluated using graded intravenous infusions of two drugs, phenylephrine and dobutamine, and by measuring the resultant cardiovascular responses. Phenylephrine and dobutamine are synthetic catecholamines, analogues of endogenous chemical messenger substances released by sympathetic nerve fibers and by adrenal medulla during stress response activation. Phenylephrine is an alpha-adrenergic agonist that increases blood pressure by constricting peripheral blood vessels. Dobutamine is beta-adrenergic agonist that stimulates myocardium to increase force of contraction and cardiac output. Stimulus-response curves for vasoconstrictor and inotropic adrenergic receptor mechanisms are constructed, from which measures of vasomotor and cardiac function, and autonomic reflex mechanisms are derived.

Clinical Relevance: Our research has suggested that there is a biomedical marker in Gulf veterans with illnesses characterized by severe unexplained chronic fatigue -- a diminished cardiovascular reactivity to cognitive stressors. Although this problem was served in all veterans with fatiguing illness, it was worst in the subset of those veterans who also had PTSD. Our data also suggested that the markedly diminished cardiovascular response to stress exhibited by this group may contribute to their functional impairment. The present investigation will determine (1) whether this impairment is due to PTSD, to the medical disorder of unexplained severe fatigue, or to an interaction between the two diagnoses, and (2) where in the system of blood pressure regulation lies the cause of abnormal stress responses. This work, therefore, may lead to better understanding of the causes of Gulf War Illnesses as well as ways to treat them.

ELIGIBILITY:
* All former military personnel who participated in the Gulf War campaign and who meet the criteria for inclusion will be eligible to participate in the study.
* Subjects with medical conditions that could explain their symptoms or with CDC-defined psychiatric exclusions (schizophrenia, mania, bulimia, and substance abuse disorders) will not participate in the study.
* Other exclusions will be pregnancy, traumatic brain injury, or a history of any form of cardiovascular disease or related symptoms.
* Other restrictions on participation will include any medication that impact on cardiovascular autonomic control, benzodiazepines, and antibiotics.
* Subjects taking nonsteroidal anti-inflammatory/analgesic agents, mild short-acting hypnotics, and SSRIs will be accepted into the study, but will be requested to withdraw from their medications with the agreement and under the supervision of their physician. These subjects will be scheduled for the study after a washout period of 5 half-lives.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf War Research Center, East Orange, New Jersey, United States